CLINICAL TRIAL: NCT00175565
Title: Effects of Fluticasone On Systemic Markers of Inflammation in Chronic Obstructive Pulmonary Disease
Brief Title: Inhaled Steroid Reduces Systemic Inflammation in COPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4027
Record Dates: First submitted 2005-09-11; First posted 2005-09-15 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema; Chronic Bronchitis
Keywords: inflammation; trial; fluticasone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic; Inflammation

INTERVENTIONS:
Drug: inhaled fluticasone 500 mcg b.i.d.

SUMMARY:
Systemic inflammation is present in chronic obstructive pulmonary disease (COPD), which has been linked to cardiovascular morbidity and mortality. We determined the effects of oral and inhaled corticosteroids on serum markers of inflammation in patients with stable COPD.

DETAILED DESCRIPTION:
We recruited patients aged 45 to 80 years, who had stable symptoms of COPD in the previous 3 months before study entry. All patients had a forced expiratory volume in one second (FEV1) after bronchodilation with 400 mcg salbutamol that was 25 to 90% of predicted, a change of less than 20% of predicted FEV1, 30 minutes following bronchodilation, and a FEV1/forced vital capacity (FVC) of less than 75%. Patients also had a history of at least 10 pack-years of smoking or prolonged exposure (>10 years) to noxious gases (e.g. diesel fumes).

At the first visit, patients, who were taking inhaled corticosteroids, were asked to immediately discontinue the use of these medications. They were allowed to take other anti-COPD medications. None of the patients took theophyllines at the time of study entry and no new medications were commenced between the first and second visits. The patients returned 4 weeks later for a second visit, at which point, they were randomized into one of the three arms of the trial: placebo capsules and a placebo puffer, fluticasone (500 mcg twice daily) and placebo capsules, or prednisone (30 mg once daily) and a placebo puffer. The trial period lasted 2 weeks. Patients were then assigned to fluticasone (500 mcg twice daily) for 8 weeks in an un-blinded fashion, followed by an additional 8 weeks of fluticasone at 1000 mcg twice daily. At each visit, we measure the participants' serum C-reactive protein (CRP) level using nephelometry in accordance with recommendations from Center for Disease Control and the American Heart Association. We also measured serum concentrations of interleukin-6 (IL-6) and monocyte chemoattractant protein-1 (MCP-1). IL-6 was measured because it is a powerful signaling cytokine for CRP expression by the liver and is a known, independent risk factor for cardiovascular events.22,23 MCP-1 was measured because it may play a central role in the pathogenesis of COPD24 and by itself is a known risk factor for atherosclerosis, myocardial infarction and cardiac deaths. All samples were analyzed in duplicate.

For analytic purposes, continuous variables that were not normally distributed (including CRP values) were log-transformed to achieve normality. We used a paired t-test to compare the log-transformed CRP values between visit 2 (i.e. at the time of randomization) and visit 3 (at the end of the randomized trial phase) within each treatment group. Similarly, using visit 2 as the referent CRP value, we used paired t-tests to compare log-transformed CRP values across the visits. To assess whether there was a gradient in the log-transformed CRP values between placebo, fluticasone and prednisone groups, we also used a Mantel-Haenszel test for trend. We reasoned a priori that oral prednisone, a more potent systemic corticosteroid than inhaled fluticasone, would have the largest effect on CRP, followed by fluticasone. Linear regression was used to examine the association between changes in interleukin-6 and log-transformed CRP values between visit 1 and 2 and between visit 2 and 3. Continuous variables are expressed as meanSD, unless otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

* stable symptoms of COPD in the previous 3 months before study entry; forced expiratory volume in one second (FEV1) after bronchodilation with 400 mcg salbutamol that was 25 to 90% of predicted, a change of less than 20% of predicted FEV1, 30 minutes following bronchodilation, and a FEV1/forced vital capacity (FVC) of less than 75%; history of at least 10 pack-years of smoking or prolonged exposure (>10 years) to noxious gases (e.g. diesel fumes).

Exclusion Criteria:

* active malignancy; unable to follow instructions; patients taking any anti-inflammatory medications

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-01; Study Completion 2003-07

PRIMARY OUTCOMES:
Change in serum C-reactive protein (CRP) levels

SECONDARY OUTCOMES:
Change in serum interleukin-6 and monocyte chemoattractant protein-1 levels

CONTACTS AND LOCATIONS:
Overall Officials: Paul Man, MD, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia

REFERENCES:
- [Result] Sin DD, Lacy P, York E, Man SF. Effects of fluticasone on systemic markers of inflammation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2004 Oct 1;170(7):760-5. doi: 10.1164/rccm.200404-543OC. Epub 2004 Jun 30. PMID 15229100
- [Result] Man SF, Sin DD. Effects of corticosteroids on systemic inflammation in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2005;2(1):78-82. doi: 10.1513/pats.200406-034MS. PMID 16113473